CLINICAL TRIAL: NCT06504329
Title: Clinical Outcomes of Enamel Matrix Derivative and Connective Tissue Graft in Modified Coronally Advanced Tunnel: A Randomized Controlled Trial
Brief Title: Clinical Outcomes of Enamel Matrix Derivative and Connective Tissue Graft in Modified Coronally Advanced Tunnel (MCAT)
Acronym: MCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Altıparmak, DDS, Research Assistant in the Department of Periodontology, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCAT - microsurgery
Record Dates: First submitted 2024-07-01; First posted 2024-07-16 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gingival Recession
Keywords: Gingival recession; modified coronally advanced tunnel; enamel matrix derivative; subepithelial connective tissue graft
MeSH Terms: conditions — Gingival Recession | interventions — Acyl-Carrier Protein S-Malonyltransferase

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Modified Coronally Advanced Tunnel (MCAT) + Subepithelial Connective Tissue Graft (SCTG) (Experimental): Participants in this arm receive the modified coronally advanced tunnel (MCAT) technique in combination with a subepithelial connective tissue graft (SCTG).
  Interventions: Procedure: Modified Coronally Advanced Tunnel (MCAT) + Subepithelial Connective Tissue Graft (SCTG)
- Modified Coronally Advanced Tunnel (MCAT) + Enamel Matrix Derivative (EMD) (Experimental): Participants in this arm receive the modified coronally advanced tunnel (MCAT) technique along with application of Emdogain (0.15 ml gel form), used as an enamel matrix derivative (EMD) to promote periodontal tissue regeneration.
  Interventions: Procedure: Modified Coronally Advanced Tunnel (MCAT) + Enamel Matrix Derivative (EMD)
- MCAT + Subepithelial Connective Tissue Graft (SCTG) + Enamel Matrix Derivative (EMD) (Experimental): Participants in this arm receive the modified coronally advanced tunnel (MCAT) technique in combination with a subepithelial connective tissue graft and application of an enamel matrix derivative (EMD; Emdogain, 0.15 ml gel form) to support periodontal tissue regeneration.
  Interventions: Procedure: Modified Coronally Advanced Tunnel (MCAT) + Subepithelial Connective Tissue Graft (SCTG); Procedure: Modified Coronally Advanced Tunnel (MCAT) + Enamel Matrix Derivative (EMD)

INTERVENTIONS:
Procedure: Modified Coronally Advanced Tunnel (MCAT) + Subepithelial Connective Tissue Graft (SCTG) — The modified coronally advanced tunnel (MCAT) technique is performed to prepare a recipient site. A subepithelial connective tissue graft (SCTG), harvested from the palate, is inserted into the tunnel using guiding sutures and stabilized. The flap is advanced coronally to completely cover the graft and achieve primary closure.
  Arms: MCAT + Subepithelial Connective Tissue Graft (SCTG) + Enamel Matrix Derivative (EMD); Modified Coronally Advanced Tunnel (MCAT) + Subepithelial Connective Tissue Graft (SCTG)
Procedure: Modified Coronally Advanced Tunnel (MCAT) + Enamel Matrix Derivative (EMD) — This intervention involves the application of enamel matrix derivative (EMD; Emdogain, 0.15 ml gel form) in conjunction with the modified coronally advanced tunnel (MCAT) technique. Following tunnel preparation, EMD is applied to the exposed root surface to enhance periodontal tissue regeneration.
  Arms: MCAT + Subepithelial Connective Tissue Graft (SCTG) + Enamel Matrix Derivative (EMD); Modified Coronally Advanced Tunnel (MCAT) + Enamel Matrix Derivative (EMD)

SUMMARY:
This study investigates the treatment of gingival recession (specifically Miller Class I and II defects) using a minimally invasive surgical approach known as the modified coronally advanced tunnel (MCAT) technique. Participants are allocated into three groups: one receiving subepithelial connective tissue grafts (SCTG), another treated with enamel matrix derivatives (EMD), and a third group receiving a combination of SCTG and EMD.

The primary objective is to evaluate the clinical effectiveness of each treatment modality in terms of root coverage, esthetic outcomes, and postoperative patient comfort. The study also aims to determine whether the combined use of SCTG and EMD provides superior clinical results compared to their individual application. Both short-term and long-term treatment outcomes are assessed to identify the most effective approach for managing gingival recession.

DETAILED DESCRIPTION:
This randomized controlled clinical trial aims to evaluate both the short- and long-term clinical outcomes of the modified coronally advanced tunnel (MCAT) technique combined with various biomaterials in the treatment of Miller Class I and II gingival recession defects.

A total of 60 systemically healthy individuals, aged between 18 and 60 years, presenting to the Department of Periodontology at Necmettin Erbakan University Faculty of Dentistry with gingival recession complaints will be included. Prior to enrollment, all participants will undergo routine periodontal examinations and nonsurgical Phase I therapy. Standard mucogingival procedures are routinely performed at this institution.

Participants will be randomly assigned to one of the following three treatment groups (n=20 each):

Group 1: MCAT + subepithelial connective tissue graft (SCTG) Group 2: MCAT + enamel matrix derivative (EMD) Group 3: MCAT + SCTG + EMD Clinical Evaluations

Clinical assessments will be conducted at baseline, 3 months, and 6 months postoperatively and will include the following parameters:

Plaque Index (PI): Assessed according to Silness and Löe (1964). Gingival Index (GI): Assessed according to Löe and Silness (1963). Gingival Recession Width (GRW): Measured horizontally at the widest point. Gingival Recession Height (GRH): Measured from the cementoenamel junction (CEJ) to the gingival margin. Keratinized Tissue Width (KTW): Measured from the gingival margin to the mucogingival junction. Probing Depth (PD) and Clinical Attachment Level (CAL): Measured at baseline and 6 months.

PD is recorded from the gingival margin to the apical extent of the sulcus; CAL is measured from the CEJ to the base of the sulcus. Intraoral Photographs: Captured at all evaluation time points. Gingival thickness will be assessed under topical anesthesia at the mid-buccal aspect, 2 mm apical to the gingival margin, using an endodontic file fitted with a rubber stopper. The distance from the file tip to the stopper will be recorded using a digital caliper.

The percentage of root coverage will be calculated based on clinical measurements, following the standardized formula described by Al-Hamdan et al. (2003).

Wound Healing Evaluation:

Sutures will be removed on postoperative day 14. Wound healing will be assessed individually for each treated site using the wound healing index proposed by Huang et al. (2005).

This study aims to provide comprehensive insights into the clinical effectiveness, esthetic outcomes, and patient-reported comfort associated with the MCAT technique when used alone or in combination with SCTG and/or EMD for the treatment of gingival recession defects.

ELIGIBILITY:
Inclusion Criteria:

Adults aged between 18 and 60 years

Systemically and periodontally healthy individuals

Non-smokers

Presence of a clearly detectable cementoenamel junction (CEJ)

No prior surgical intervention at the selected sites

No periodontal pockets deeper than 3 mm

No signs of occlusal trauma

Exclusion Criteria:

Pregnancy or lactation

Use of antibiotics in the past 6 months

Presence of any systemic condition that may contraindicate periodontal surgery, including:

Diabetes mellitus

Impaired glucose tolerance

Endocrine disorders

Cardiovascular diseases

Declined to participate or failed to meet inclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Root Surface Coverage (%RC) | 6 months postoperatively
  The percentage of root surface coverage will be calculated based on changes in the exposed root surface area before and after treatment. The exposed area is estimated by multiplying the height and width of the gingival recession. The difference between the baseline and 6-month postoperative values will be used to determine the percentage of coverage. Results will be expressed as a percentage (%). This approach reflects the clinical effectiveness of the intervention and is based on the method described by Al-Hamdan et al. (2003).

SECONDARY OUTCOMES:
Gingival Index (GI) | Baseline, 1, 3, and 6 months postoperatively
  Gingival inflammation will be scored using the Löe and Silness Gingival Index (1963), with scores ranging from 0 (normal) to 3 (severe inflammation).
Plaque Index (PI) | Baseline, 1, 3, and 6 months postoperatively.
  Oral hygiene will be assessed using the Silness and Löe Plaque Index (1964), scored from 0 (no plaque) to 3 (abundant plaque accumulation).
Gingival Recession Height (GRH) | Baseline, 1, 3, and 6 months postoperatively
  Gingival recession height will be measured in millimeters from the cementoenamel junction (CEJ) to the gingival margin using a periodontal probe.
Gingival Recession Width (GRW) | Baseline, 1, 3, and 6 months postoperatively.
  Gingival recession width will be measured in millimeters as the horizontal distance between the mesial and distal borders of the recession at its widest point. A periodontal probe will be positioned parallel to the cementoenamel junction to record the measurement.
Clinical Attachment Level (CAL) | Baseline and 6 months postoperatively.
  Clinical attachment level will be measured in millimeters as the distance from the cementoenamel junction (CEJ) to the base of the sulcus using a periodontal probe at the mid-vestibular aspect of the tooth.
Keratinized Tissue Width (KTW) | Baseline, 1, 3, and 6 months postoperatively.
  Keratinized tissue width (in millimeters) will be measured from the free gingival margin to the mucogingival junction using a periodontal probe. Measurements will be taken at the mid-point of the recession site.
Gingival Thickness | Baseline and 6 months postoperatively.
  Gingival thickness (in millimeters) will be measured at the mid-buccal region, 2 mm apical to the gingival margin, under topical anesthesia. A #25 endodontic spreader with a rubber stopper will be inserted perpendicular to the gingival surface until contact with hard tissue is achieved. The distance from the tip to the stopper will be recorded using a digital caliper.
Wound Healing Index (WHI) | 2 weeks postoperatively.
  ound healing will be assessed two weeks postoperatively upon suture removal, using the Wound Healing Index (WHI) as defined by Huang et al. (2005). Each surgical site will be scored as follows:
  Score 1: Uneventful healing without gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence.
  Score 2: Slight edema, erythema, patient discomfort, or flap dehiscence, but without suppuration or infection.
  Score 3: Poor healing with significant edema, erythema, patient discomfort, flap dehiscence, or presence of infection.
Probing Depth (PD) | Baseline and 6 months postoperatively.
  Probing depth will be measured using a Williams periodontal probe (Hu-Friedy) at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual), parallel to the tooth's long axis. The probe will be inserted with gentle pressure (~0.25 N) until slight resistance is felt at the base of the sulcus. The distance from the free gingival margin to the base of the pocket will be recorded in millimeters and rounded to the nearest whole number.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No